CLINICAL TRIAL: NCT02053142
Title: Prospective Study of Pharmacokinetics, Clinical and Virologic Response to Acyclovir Episodic Therapy for Genital Herpes Ulcers in HIV Negative African Women
Brief Title: Acyclovir Therapy for Genital Herpes Ulcers in HIV Negative African Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIDRZ 1208/IRB12-0390
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2014-12

CONDITIONS: Ulcers of Female Genital Organs
Keywords: Pharmacokinetics; Herpes simplex virus; Genital herpes ulcers
MeSH Terms: conditions — Herpes Simplex | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 PK (Experimental): 400mg dose of acyclovir taken orally, followed by 2 ml blood plasma collection at 1,2,4,6 and 8 hours.
  Interventions: Drug: Acyclovir
- Acyclovir (Active Comparator): 400 mg Acyclovir three times daily for 5 days
  Interventions: Drug: Acyclovir
- Placebo (Placebo Comparator): Placebo three times daily for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acyclovir — Single dose of acyclovir 200mg was given for pk study
  Arms: Acyclovir; Part 1 PK
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a prospective study to evaluate the pharmacokinetics, clinical and virologic response to acyclovir episodic therapy for genital herpes ulcers in HIV negative African women.

DETAILED DESCRIPTION:
This is a two-part study designed to measure the Area Under the Curve (AUC) from a single dose of acyclovir 400mg in 60 African HIV-negative heterosexual women who have a history of genital ulcer disease (GUD), are HSV-2 seropositive and HIV-1 seronegative. The study will also examine the time to healing of genital lesion and duration of HSV shedding from GUD among 90 HIV negative African women who have a history of GUD and are Herpes Simplex Virus (HSV)-2 seropositive and HIV-1 seronegative randomized in a 2:1 ratio to receive episodic acyclovir or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative as determined by concordant rapid testing
* HSV-2 seropositive (Focus HerpeSelect EIA >3.4)
* At least one prior occurrence of GUD
* 18 to 50 years of age

Exclusion Criteria:

* Current use, or use within the past 7 days, of acyclovir, valacyclovir, or famciclovir
* Prior hypersensitivity and/or allergic reaction to acyclovir
* Use of probenecid, which prolongs renal excretion of acyclovir
* Current use, or use within the past 28 days, of an investigational agent
* Currently pregnant or nursing
* Currently plan to become pregnant during the next 3 months
* Currently consume, on average, more than 7 drinks of alcohol per week (for Part I)
* Current use of more than 20 cigarettes daily (for Part I)
* Any condition that in the opinion of the investigator will interfere with successful completion of all study procedures.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (AUC) | 0, 2, 3, 4, 6 and 8 hours post acyclovir administration
  Blood will be drawn for pharmacokinetic measures to determine whether there is a difference in African women vs. the existing AUC data for women and men in North America and Europe.

SECONDARY OUTCOMES:
Time to re-epithelization and time to cessation of HSV shedding | days 1-5, 7, 9, 11 and 13
  Daily assessment of response of genital lesions over 13 days by time to healing and duration of HSV shedding during acyclovir 400mg orally three times daily versus placebo three times daily for 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Reid, MD, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Reichman RC, Badger GJ, Mertz GJ, Corey L, Richman DD, Connor JD, Redfield D, Savoia MC, Oxman MN, Bryson Y, et al. Treatment of recurrent genital herpes simplex infections with oral acyclovir. A controlled trial. JAMA. 1984 Apr 27;251(16):2103-7. PMID 6368877
- [Background] Nilsen AE, Aasen T, Halsos AM, Kinge BR, Tjotta EA, Wikstrom K, Fiddian AP. Efficacy of oral acyclovir in the treatment of initial and recurrent genital herpes. Lancet. 1982 Sep 11;2(8298):571-3. doi: 10.1016/s0140-6736(82)90658-4. PMID 6125728
- [Background] Celum, C., et al., HSV-2 Suppressive Therapy for Prevention of HIV Acquisition: Results of HPTN 039. The Lancet, in press.
- [Background] Reitano M, Tyring S, Lang W, Thoming C, Worm AM, Borelli S, Chambers LO, Robinson JM, Corey L. Valaciclovir for the suppression of recurrent genital herpes simplex virus infection: a large-scale dose range-finding study. International Valaciclovir HSV Study Group. J Infect Dis. 1998 Sep;178(3):603-10. doi: 10.1086/515385. PMID 9728526
- [Background] Gupta R, Wald A, Krantz E, Selke S, Warren T, Vargas-Cortes M, Miller G, Corey L. Valacyclovir and acyclovir for suppression of shedding of herpes simplex virus in the genital tract. J Infect Dis. 2004 Oct 15;190(8):1374-81. doi: 10.1086/424519. Epub 2004 Sep 20. PMID 15378428
- [Background] Watson-Jones D, Weiss HA, Rusizoka M, Changalucha J, Baisley K, Mugeye K, Tanton C, Ross D, Everett D, Clayton T, Balira R, Knight L, Hambleton I, Le Goff J, Belec L, Hayes R; HSV trial team; Steering and Data Monitoring Committees. Effect of herpes simplex suppression on incidence of HIV among women in Tanzania. N Engl J Med. 2008 Apr 10;358(15):1560-71. doi: 10.1056/NEJMoa0800260. Epub 2008 Mar 12. PMID 18337596
- [Background] Blum, M., et al., The bioavailability and pharmacokinetics of ZOVIRAX 200 mg capsules vs solution in normal volunteers at risk of developing herpes simplex virus infections (Protocol P12-83). Burroughs Wellcome Document No. TEIN/82/0001.
- [Background] De Miranda, P. and D. Page, Systemic absorption and pharmacokinetics of acyclovir (ZOVIRAX) when administered orally in multiple doses of 600 mg to immunocompromised patients with herpes infections (Protocol 12-30, Dr. R. Whitley). Burroughs Wellcome Document No. TEIN/82/0007.
- [Background] De Miranda, P. and D. Page, Systemic absorption and pharmacokinetics of acyclovir (ZOVIRAX) when administered orally in multiple doses of 800 mg to immunocompromised patients with herpes infections (Protocol 12-30, Dr. R. Whitley) Burroughs Wellcome Document No. TEIN/83/0001.
- [Background] Blum, M. and S. Liao, Pharmacokinetics and relative bioavailability of acyclovir capsules (ZOVIRAX) after multiple oral doses (Interim summary of study P12-32) amendment). Burroughs Wellcome Document No. TYBH/83/0001.
- [Background] Amini H, Javan M, Gazerani P, Ghaffari A, Ahmadiani A. Lack of bioequivalence between two aciclovir tablets in healthy subjects. Clin Drug Investig. 2008;28(1):47-53. doi: 10.2165/00044011-200828010-00006. PMID 18081360
- [Background] Bahrami G, Mirzaeei Sh, Kiani A. Determination of acyclovir in human serum by high-performance liquid chromatography using liquid-liquid extraction and its application in pharmacokinetic studies. J Chromatogr B Analyt Technol Biomed Life Sci. 2005 Feb 25;816(1-2):327-31. doi: 10.1016/j.jchromb.2004.11.038. PMID 15664366
- [Background] Palma-Aguirre JA, Absalon-Reyes JA, Novoa-Heckel G, de Lago A, Oliva I, Rodriguez Z, Gonzalez-de la Parra M, Burke-Fraga V, Namur S. Bioavailability of two oral suspension and two oral tablet formulations of acyclovir 400 mg: two single-dose, open-label, randomized, two-period crossover comparisons in healthy Mexican adult subjects. Clin Ther. 2007 Jun;29(6):1146-52. doi: 10.1016/j.clinthera.2007.06.007. PMID 17692728
- [Background] Vergin H, Kikuta C, Mascher H, Metz R. Pharmacokinetics and bioavailability of different formulations of aciclovir. Arzneimittelforschung. 1995 Apr;45(4):508-15. PMID 7779152
- [Background] Landowski CP, Sun D, Foster DR, Menon SS, Barnett JL, Welage LS, Ramachandran C, Amidon GL. Gene expression in the human intestine and correlation with oral valacyclovir pharmacokinetic parameters. J Pharmacol Exp Ther. 2003 Aug;306(2):778-86. doi: 10.1124/jpet.103.051011. Epub 2003 May 15. PMID 12750437
- [Background] Steingrimsdottir H, Gruber A, Palm C, Grimfors G, Kalin M, Eksborg S. Bioavailability of aciclovir after oral administration of aciclovir and its prodrug valaciclovir to patients with leukopenia after chemotherapy. Antimicrob Agents Chemother. 2000 Jan;44(1):207-9. doi: 10.1128/AAC.44.1.207-209.2000. PMID 10602752
- [Background] Kimberlin DF, Weller S, Whitley RJ, Andrews WW, Hauth JC, Lakeman F, Miller G. Pharmacokinetics of oral valacyclovir and acyclovir in late pregnancy. Am J Obstet Gynecol. 1998 Oct;179(4):846-51. doi: 10.1016/s0002-9378(98)70176-0. PMID 9790357
- [Background] Frenkel LM, Brown ZA, Bryson YJ, Corey L, Unadkat JD, Hensleigh PA, Arvin AM, Prober CG, Connor JD. Pharmacokinetics of acyclovir in the term human pregnancy and neonate. Am J Obstet Gynecol. 1991 Feb;164(2):569-76. doi: 10.1016/s0002-9378(11)80023-2. PMID 1847004
- [Background] Haddad J, Langer B, Astruc D, Messer J, Lokiec F. Oral acyclovir and recurrent genital herpes during late pregnancy. Obstet Gynecol. 1993 Jul;82(1):102-4. PMID 8390630
- [Background] Stone KM, Whittington WL. Treatment of genital herpes. Rev Infect Dis. 1990 Jul-Aug;12 Suppl 6:S610-9. doi: 10.1093/clinids/12.supplement_6.s610. PMID 2166968
- [Background] Spruance SL, Jones TM, Blatter MM, Vargas-Cortes M, Barber J, Hill J, Goldstein D, Schultz M. High-dose, short-duration, early valacyclovir therapy for episodic treatment of cold sores: results of two randomized, placebo-controlled, multicenter studies. Antimicrob Agents Chemother. 2003 Mar;47(3):1072-80. doi: 10.1128/AAC.47.3.1072-1080.2003. PMID 12604544
- [Background] Bodsworth NJ, Crooks RJ, Borelli S, Vejlsgaard G, Paavonen J, Worm AM, Uexkull N, Esmann J, Strand A, Ingamells AJ, Gibb A. Valaciclovir versus aciclovir in patient initiated treatment of recurrent genital herpes: a randomised, double blind clinical trial. International Valaciclovir HSV Study Group. Genitourin Med. 1997 Apr;73(2):110-6. doi: 10.1136/sti.73.2.110. PMID 9215092
- [Background] Sacks SL, Aoki FY, Diaz-Mitoma F, Sellors J, Shafran SD. Patient-initiated, twice-daily oral famciclovir for early recurrent genital herpes. A randomized, double-blind multicenter trial. Canadian Famciclovir Study Group. JAMA. 1996 Jul 3;276(1):44-9. PMID 8667538
- [Background] Spruance SL, Tyring SK, DeGregorio B, Miller C, Beutner K. A large-scale, placebo-controlled, dose-ranging trial of peroral valaciclovir for episodic treatment of recurrent herpes genitalis. Valaciclovir HSV Study Group. Arch Intern Med. 1996 Aug 12-26;156(15):1729-35. PMID 8694673
- [Background] Aoki FY, Tyring S, Diaz-Mitoma F, Gross G, Gao J, Hamed K. Single-day, patient-initiated famciclovir therapy for recurrent genital herpes: a randomized, double-blind, placebo-controlled trial. Clin Infect Dis. 2006 Jan 1;42(1):8-13. doi: 10.1086/498521. Epub 2005 Nov 23. PMID 16323085
- [Background] Wald A, Carrell D, Remington M, Kexel E, Zeh J, Corey L. Two-day regimen of acyclovir for treatment of recurrent genital herpes simplex virus type 2 infection. Clin Infect Dis. 2002 Apr 1;34(7):944-8. doi: 10.1086/339325. Epub 2002 Feb 20. PMID 11880960
- [Background] Leone PA, Trottier S, Miller JM. Valacyclovir for episodic treatment of genital herpes: a shorter 3-day treatment course compared with 5-day treatment. Clin Infect Dis. 2002 Apr 1;34(7):958-62. doi: 10.1086/339326. Epub 2002 Feb 20. PMID 11880962
- [Background] Wald A, Huang ML, Carrell D, Selke S, Corey L. Polymerase chain reaction for detection of herpes simplex virus (HSV) DNA on mucosal surfaces: comparison with HSV isolation in cell culture. J Infect Dis. 2003 Nov 1;188(9):1345-51. doi: 10.1086/379043. Epub 2003 Oct 31. PMID 14593592
- [Background] Wald A, Zeh J, Selke S, Warren T, Ryncarz AJ, Ashley R, Krieger JN, Corey L. Reactivation of genital herpes simplex virus type 2 infection in asymptomatic seropositive persons. N Engl J Med. 2000 Mar 23;342(12):844-50. doi: 10.1056/NEJM200003233421203. PMID 10727588
- [Background] Diaz-Mitoma F, Ruben M, Sacks S, MacPherson P, Caissie G. Detection of viral DNA to evaluate outcome of antiviral treatment of patients with recurrent genital herpes. J Clin Microbiol. 1996 Mar;34(3):657-63. doi: 10.1128/jcm.34.3.657-663.1996. PMID 8904433
- [Background] Leone P, Warren T, Hamed K, Fife K, Wald A. Famciclovir reduces viral mucosal shedding in HSV-seropositive persons. Sex Transm Dis. 2007 Nov;34(11):900-7. doi: 10.1097/OLQ.0b013e318063c749. PMID 17538513
- [Background] Bavaro JB, Drolette L, Koelle DM, Almekinder J, Warren T, Tyring S, Wald A. One-day regimen of valacyclovir for treatment of recurrent genital herpes simplex virus 2 infection. Sex Transm Dis. 2008 Apr;35(4):383-6. doi: 10.1097/OLQ.0b013e31815e4190. PMID 18362859
- [Background] Goldberg LH, Kaufman R, Conant MA, Sperber J, Allen ML, Illeman M, Chapman S. Oral acyclovir for episodic treatment of recurrent genital herpes. Efficacy and safety. J Am Acad Dermatol. 1986 Aug;15(2 Pt 1):256-64. doi: 10.1016/s0190-9622(86)70165-5. PMID 3745529
- [Background] Tyring SK, Douglas JM Jr, Corey L, Spruance SL, Esmann J. A randomized, placebo-controlled comparison of oral valacyclovir and acyclovir in immunocompetent patients with recurrent genital herpes infections. The Valaciclovir International Study Group. Arch Dermatol. 1998 Feb;134(2):185-91. doi: 10.1001/archderm.134.2.185. PMID 9487210
- [Background] Freeman EE, Weiss HA, Glynn JR, Cross PL, Whitworth JA, Hayes RJ. Herpes simplex virus 2 infection increases HIV acquisition in men and women: systematic review and meta-analysis of longitudinal studies. AIDS. 2006 Jan 2;20(1):73-83. doi: 10.1097/01.aids.0000198081.09337.a7. PMID 16327322
- [Background] Rebbapragada A, Wachihi C, Pettengell C, Sunderji S, Huibner S, Jaoko W, Ball B, Fowke K, Mazzulli T, Plummer FA, Kaul R. Negative mucosal synergy between Herpes simplex type 2 and HIV in the female genital tract. AIDS. 2007 Mar 12;21(5):589-98. doi: 10.1097/QAD.0b013e328012b896. PMID 17314521
- [Background] Belec, L., et al. Impact of HSV-2 Episodic Therapy on HIV-1 and HSV-2 Genital Shedding and Ulcer Healing Among Women in Ghana and the Central African Republic: Randomized Double-Blind Placebo-Controlled trial. in XXth Annual Conference of the International Union Against STI. 2006. Versailles, France.
- [Background] Paz-Bailey, G., et al. Impact of Episodic Acyclovir Therapy on Genital Ulcer Duration and HIV Shedding from Herpetic Ulcers Among Men in South Africa. in 17th International Society for STD Research Meeting. 2007. Seattle, Washington, USA.
- See also: University of North Carolina website — http://www.unc.edu